CLINICAL TRIAL: NCT05391594
Title: Effect of Optimal Trunk Support on Academic Engagement of Children With Moderate to Severe Disability
Brief Title: Effect of Trunk Support on Academic Engagement of Children With Severe Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO18010001
Record Dates: First submitted 2018-11-26; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Cerebral Palsy; Traumatic Brain Injury; Metabolic Disease; Hypotonia
Keywords: posture; trunk control; assistive device
MeSH Terms: conditions — Cerebral Palsy; Brain Injuries, Traumatic; Metabolic Diseases; Muscle Hypotonia

STUDY DESIGN:
Intervention Model Description: Single Subject Research Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single Subject Design (Experimental): The investigators will use a longitudinal design with baseline, immediate and post-intervention data collections. The intervention will include customized posture support in seated, standing or walking devices that will be used in the child's educational setting or home (for early intervention) to facilitate specific educational activities.
  Interventions: Device: customized posture support

INTERVENTIONS:
Device: customized posture support — We will provide customized modifications for seated or standing or walking devices based on the child's segmental level of control

SUMMARY:
This study evaluates the effect of optimizing trunk support based on segmental principles of trunk control, on academic engagement of children in academic settings.

DETAILED DESCRIPTION:
Head and trunk posture control are foundational skills, impacting vision, communication, swallowing, eating, reaching, and gait. Vision, communication and upper extremity skills are critical for participation in educational settings. From an academic point of view, participants with poor trunk stability have difficulties staying erect and keeping their head and trunk steady. This interferes with concentration, reduces ability and aptitude for learning and can lead to fatigue and reduced time on task. Examination of the effect of optimal trunk support may yield critical information regarding academic engagement in children with moderate to severe disability.

The investigators propose to facilitate use of a segmental approach by physical and occupational therapists in educational settings. Activities will include identifying level of trunk control and applying segmental principles to adapt participant's positioning devices for optimal function.

ELIGIBILITY:
Inclusion Criteria:

* Referral from physical, occupational or speech therapist working in Hartford Public School District or Connecticut Birth to Three,
* Segmental deficit in trunk control as measured by Segmental Assessment of Trunk Control
* parent or guardian consent that includes permission for video data collection and sharing of IEP (individualized education plan) or IFSP (individualized family support plan).

Exclusion Criteria:

* pain that interferes with positioning,
* impending surgery that will result in extended absence from school

Ages: 3 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Video Behavior Coding of time "on task" for selected IEP or IFSP goals. | On day 1 and one additional date at least 3 weeks later.
  Frequency and duration of 'on task' behavior will be coded for 2 or 3 of the child's existing education goals under two conditions, when child is in usual positioning equipment and in segmentally optimized equipment. Goals of interest reflect motor behaviors that promote task performance or interaction. These include 1) eye gaze (at people or objects), 2) reaching, 3) object manipulation, 4) head turning and 5) making choices (using eye gaze or reach).

SECONDARY OUTCOMES:
Change in vertical alignment of head | On the day 1 and one additional date at least 3 weeks later.
  frequency and duration of upright 'head position' will be coded for 2 or 3 of the child's existing education goals under two conditions, when child is in usual positioning equipment and in segmentally optimized equipment.
parent, teacher or aide device use record | from day 1 to second session at least 3 weeks later)
  frequency and duration of device use and comments about child and teachers response to using the device.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Saavedra, Principal Investigator — University of Hartford
Locations (3):
- United States (3):
  - Children's Therapy Services, Connecticut Birth to Three, Cheshire, Connecticut
  - Hartford Public Schools, Hartford, Connecticut
  - CREC, Connecticut Birth to Three, Wethersfield, Connecticut